CLINICAL TRIAL: NCT02826122
Title: Prevalence of Diastolic Dysfunction and Effects of Conservative Lifestyle Treatment in Patients With Morbid Obesity
Brief Title: Diastolic Dysfunction During Conservative Lifestyle Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: LHL Helse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/833
Record Dates: First submitted 2016-07-05; First posted 2016-07-07 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FitBit APP (Active Comparator): FitBit Zip APP registers and give feed-back on number of steps per day, distance and calories burned.
  Interventions: Device: FitBit APP
- Pai APP (Experimental): Mio Pai APP registers duration and intensity of the Activity and give feed back as activity Points.
  Interventions: Device: Pai APP

INTERVENTIONS:
Device: Pai APP — Prescription: Target 100 PAI Points per week
  Other Names: Personal Activity Intelligence (PAI) application; MIO Fuse Wristband
  Arms: Pai APP
Device: FitBit APP — Prescription: Target daily 10.000 steps
  Other Names: FitBit Zip
  Arms: FitBit APP

SUMMARY:
The Purpose of this study is to 1) investigate prevalence of diastolic dysfunction in patients with morbid obesity attending a conservative lifestyle change program, 2) investigate effects on cardiac function, cardiorespiratory Fitness, body composition, quality of life and cardiovascular risk through the program, 3) investigate feasibility of introducing two different activity monitors throughout the program, and 4) comparing compliance to activity sensor market leader FitBit Application versus Mio Pai Application

ELIGIBILITY:
Inclusion Criteria:

* BMI > 40 kg/m2 (or BMI > 35 kg/m2 with comorbidity)
* Stable weight last Three months (≤ 2 kg variation)
* Norwegian speaking
* Smartphone

Exclusion Criteria:

* Other weight reduction treatment, including medication affecting appetite
* Known chronic cardiac condition
* Previous bariatric surgery
* Alcohol or other substitute abuse
* Psychiatric disorder needing treatment, including eating disorders
* Pregnancy or planned pregnancy during project period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
diastolic dysfunction | 18 months
  echocardiac examination at baseline assessed by GE Healthcare Vivid E9, Horten, Norway

SECONDARY OUTCOMES:
diastolic function | 4 months
  echocardiac examination assessed by GE Healthcare Vivid E9, Horten, Norway
diastolic function | 12 months
  echocardiac examination assessed by GE Healthcare Vivid E9, Horten, Norway
Cardiorespiratory fitness | 4 months
  Peak oxygen uptake assessed by Jaeger oxycon pro; Erich Jaeger GmbH, Hoechberg, Germany
Cardiorespiratory fitness | 12 months
  Peak oxygen uptake assessed by Jaeger oxycon pro; Erich Jaeger GmbH, Hoechberg, Germany
Cardiorespiratory fitness | 18 months
  Peak oxygen uptake assessed by Jaeger oxycon pro; Erich Jaeger GmbH, Hoechberg, Germany
Body composition | 4 months
  Body composition assessed by bioelectrical impedance (instrument InBody 770, produced by BIOSPACE, Seoul, Korea)
Body composition | 12 months
  Body composition assessed by bioelectrical impedance (instrument InBody 770, produced by BIOSPACE, Seoul, Korea)
Body composition | 18 months
  Body composition assessed by bioelectrical impedance (instrument InBody 770, produced by BIOSPACE, Seoul, Korea)
Body Mass Index | 4 months
  Weight derived by squared height
Body Mass Index | 12 months
  Weight derived by squared height
Body Mass Index | 18 months
  Weight derived by squared height
Waist line | 4 months
  tape measure in centimeters
Waist line | 12 months
  tape measure in centimeters
Waist line | 18 months
  tape measure in centimeters
Physical Activity Questionnaire | 4 months
  HUNT 1 physical activity questionnaire
Physical Activity Questionnaire | 12 months
  HUNT 1 physical activity questionnaire
Physical Activity Questionnaire | 18 months
  HUNT 1 physical activity questionnaire
Quality of life | 4 months
  Impact of Weight on Quality of Life Short Form (IWQOL-Lite); Kolotkin
Quality of life | 12 months
  Impact of Weight on Quality of Life Short Form (IWQOL-Lite); Kolotkin
Quality of life | 18 months
  Impact of Weight on Quality of Life Short Form (IWQOL-Lite); Kolotkin
Symptoms of anxiety and depression | 4 months
  Hospital Anxiety and Depression Scale; Zigmond & Snaith
Symptoms of anxiety and depression | 12 months
  Hospital Anxiety and Depression Scale; Zigmond & Snaith
Symptoms of anxiety and depression | 18 months
  Hospital Anxiety and Depression Scale; Zigmond & Snaith
Glucose concentration in blood | 4 months
Glucose concentration in blood | 12 months
Glucose concentration in blood | 18 months
Glycosylated haemoglobin (HbA1c) concentration in blood | 4 months
Glycosylated haemoglobin (HbA1c) concentration in blood | 12 months
Glycosylated haemoglobin (HbA1c) concentration in blood | 18 months
LDL concentration in blood | 4 months
  Low Density Cholesterol
LDL concentration in blood | 12 months
  Low Density Cholesterol
LDL concentration in blood | 18 months
  Low Density Cholesterol
HDL concentration in blood | 4 months
  High Density Cholesterol
HDL concentration in blood | 12 months
  High Density Cholesterol
HDL concentration in blood | 18 months
  High Density Cholesterol
Concentration of total cholesterol in blood | 4 months
Concentration of total cholesterol in blood | 12 months
Concentration of total cholesterol in blood | 18 months
Concentration of triglycerides in blood serum | 4 months
Concentration of triglycerides in blood serum | 12 months
Concentration of triglycerides in blood serum | 18 months
Concentration of HS-CRP in blood serum | 4 months
  High Sensitive C-reactive protein
Concentration of HS-CRP in blood serum | 12 months
  High Sensitive C-reactive protein
Concentration of HS-CRP in blood serum | 18 months
  High Sensitive C-reactive protein
C-peptide concentration in blood | 4 months
C-peptide concentration in blood | 12 months
C-peptide concentration in blood | 18 months
Leukocyte concentration in blood | 4 months
Leukocyte concentration in blood | 12 months
Leukocyte concentration in blood | 18 months
Potassium (K) concentration in blood | 4 months
Potassium (K) concentration in blood | 12 months
Potassium (K) concentration in blood | 18 months
Sodium (Na) concentration in blood | 4 months
Sodium (Na) concentration in blood | 12 months
Sodium (Na) concentration in blood | 18 months
Creatinine concentration in blood | 4 months
Creatinine concentration in blood | 12 months
Creatinine concentration in blood | 18 months
Apo-A concentration in blood serum | 4 months
  Apolipoprotein A
Apo-A concentration in blood serum | 12 months
  Apolipoprotein A
Apo-A concentration in blood serum | 18 months
  Apolipoprotein A
Apo-B concentration in blood serum | 4 months
  Apolipoprotein B
Apo-B concentration in blood serum | 12 months
  Apolipoprotein B
Apo-B concentration in blood serum | 18 months
  Apolipoprotein B
NT-ProBNP concentration in plasma | 4 months
  N-Terminal Brain Natriuretic Peptide
NT-ProBNP concentration in plasma | 12 months
  N-Terminal Brain Natriuretic Peptide
NT-ProBNP concentration in plasma | 18 months
  N-Terminal Brain Natriuretic Peptide
Lp(a) concentration in blood serum | 4 months
  Lipoprotein(a)
Lp(a) concentration in blood serum | 12 months
  Lipoprotein(a)
Lp(a) concentration in blood serum | 18 months
  Lipoprotein(a)

OTHER OUTCOMES:
Feasibility | 4 months
  measured as attrition rate, Activity sensor errors
Feasibility | 12 months
  measured as attrition, Activity sensor errors,
Feasibility | 18 months
  measured as attrition, Activity sensor errors,
Compliance | 4 months
  actual use of Activity sensors; obtaining 80 % or more of prescribed physical Activity in home periods
Compliance | 12 months
  actual use of Activity sensors; obtaining 80 % or more of prescribed physical Activity in home periods
Compliance | 18 months
  actual use of Activity sensors; obtaining 80 % or more of prescribed physical Activity in home periods
Meal frequency, compliance With a healthier lifestyle | 4 months
  HUNT 3 questionnaire
Meal frequency, compliance With a healthier lifestyle | 12 months
  HUNT 3 questionnaire
Meal frequency, compliance With a healthier lifestyle | 18 months
  HUNT 3 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Line Oldervoll, PhD, Principal Investigator — LHL klinikkene / NTNU
Locations (1):
- LHL-Klinikkene, Røros, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Oldervoll LM, Gjestad R, Hilmarsen C C, Ose A, Gullikstad L, Wisloff U, Kulseng B, Grimsmo J. Diastolic function and cardiovascular risk among patients with severe obesity referred to a lifestyle-program - a pilot study. Scand Cardiovasc J. 2023 Dec;57(1):8-16. doi: 10.1080/14017431.2022.2146185. PMID 36404730